CLINICAL TRIAL: NCT02576184
Title: Mesh Reinforcement During Temporary Stoma Closure After Sphincter-Saving Rectal Cancer Surgery: A Randomized-controlled Trial
Brief Title: Mesh Reinforcement During Temporary Stoma Closure After Sphincter-Saving Rectal Cancer Surgery
Acronym: MEMBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P140312; 2015-A00410-49 (Other: IDRCB)
Record Dates: First submitted 2015-10-05; First posted 2015-10-15 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Incisional Hernia After Diverting Stoma Closure
Keywords: Incisional hernia; Stoma; rectal cancer; synthetic mesh; biologic mesh
MeSH Terms: conditions — Incisional Hernia; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Biologic mesh Synthetic mesh
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biologic Mesh (Experimental): Biologic mesh placed in retromuscular position
  Interventions: Device: Biologic Mesh
- Synthetic Mesh (Experimental): Synthetic mesh placed in retromuscular position
  Interventions: Device: Synthetic Mesh
- No Mesh (No Intervention): No mesh

INTERVENTIONS:
Device: Biologic Mesh — Biologic mesh placed in retromuscular position during ileostoma closure
  Arms: Biologic Mesh
Device: Synthetic Mesh — synthetic mesh placed in retromuscular position during ileostoma closure
  Arms: Synthetic Mesh

SUMMARY:
This study aim to assess long-term results of an incisional hernia-prophylactic mesh placement during stoma reversal after total mesorectal excision (TME) for rectal cancer

DETAILED DESCRIPTION:
This study aim to assess long-term results of an incisional hernia-prophylactic mesh placement during stoma reversal after TME for rectal cancer.

Patients are randomized in 3 groups : no mesh, synthetic mesh (Parietex, Covidien), biologic mesh (Cellis, Meccelis). Meshes are placed in retromuscular position after diverting ileostomy closure.

Primary endpoint is radiological incisional hernia rate, assessed on CT-scan, at the end of follow-up Secondary endpoints include postoperative morbidity, postoperative pain, postoperative quality of life, long-term clinical incisional hernia rate.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Operated on for diverting ileostoma closure after sphincter saving rectal cancer surgery, irrespective of the time delay between ileostoma closure and rectal cancer surgery
* Signed consent
* Affiliation to the French social security system

Exclusion Criteria:

* Emergency surgery
* History of laparotomy before ileostoma closure.
* Surgery associated to the ileostoma closure, excluding appendectomy or liver biopsy
* Lactating or pregnant woman
* Allergy to porcine product or collagen-based product. Allergy to polypropylene.
* Participation to another protocol focusing on ileostoma closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
radiological incisional hernia rate | up to 36 months
  Primary endpoint is radiological incisional hernia rate, assessed on CT-scan, at the end of follow-up.
  Statistical analysis will be performed as soon as follow-up reach 12 months for last included patient

SECONDARY OUTCOMES:
Postoperative morbidity | 30 days
  Postoperative morbidity
Postoperative pain | 36 months
  Score Brief Pain Inventory
Postoperative rehospitalization | 36 months
  Case report form data
Postoperative reintervention | 36 months
  Case report form data
Quality of life (The Short Form (36) Health Survey score) | 12 months
  The Short Form (36) Health Survey
Clinical incisional hernia rate | 36 months
  Clinical incisional hernia rate : Statistical analysis will be performed as soon as follow-up reach 12 months for last included patient

CONTACTS AND LOCATIONS:
Overall Officials: Leon Maggiori, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Chirurgie Colorectale - Hôpital Beaujon, Clichy, France

REFERENCES:
- [Derived] Vu BK, Lam J, Sherman MJ, Tam MS. Prophylactic Biosynthetic Retrorectus Mesh Placement During Stoma Reversal Reduces the Rate of Stoma Site Incisional Hernia. Perm J. 2024 Jun 14;28(2):16-25. doi: 10.7812/TPP/23.115. Epub 2024 Apr 23. PMID 38652519